CLINICAL TRIAL: NCT04274114
Title: Efficacy of L-glutamine for the Treatment of Generalized Anxiety Disorder: a Randomized Controlled Trial
Brief Title: Treatment of Adults With Generalized Anxiety Disorder Using Glutamine
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Inhability to recruit further participants due to SARS-CoV-2 pandemics.
Sponsor: Hospital Universitario Dr. Jose E. Gonzalez (Other)
Collaborators: Instituto de Información e Investigación en Salud Mental A. C. (Unknown)
Responsible Party: Principal Investigator, José Alfonso Ontiveros Sánchez De la Barquera, Associate Professor, Hospital Universitario Dr. Jose E. Gonzalez
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PS18-00018
Record Dates: First submitted 2020-02-14; First posted 2020-02-18 (Actual); Last update posted 2021-02-11 (Actual); Status verified 2021-02

CONDITIONS: Generalized Anxiety Disorder
Keywords: generalized anxiety disorder; randomized controlled trial; psychopharmacology; drug therapy; glutamine
MeSH Terms: conditions — Generalized Anxiety Disorder | interventions — Glutamine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Patients in this group will receive flexible doses of L-glutamine ranging from 5 to 25 grams once daily for 8 weeks. L-glutamine is administered as a powder dissolved in water.
  Interventions: Drug: L Glutamine
- Placebo group (Placebo Comparator): Patients in this group will receive flexible doses of placebo ranging from 5 to 25 grams once daily for 8 weeks. Placebo is administered as a powder dissolved in water.
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: L Glutamine — Powder
  Arms: Experimental group
Drug: Placebos — Powder
  Arms: Placebo group

SUMMARY:
The objective of this randomized clinical trial is to examine the efficacy of L-glutamine for the treatment of generalized anxiety disorder compared versus placebo.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients with generalized anxiety disorder defined by the criteria of the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-V)
* Generalized anxiety disorder is the primary psychiatric disorder.
* Untreated patients or; patients treated with paroxetine, sertraline, citalopram, escitalopram, venlafaxine or duloxetine at least for 6 weeks on a stable dose; or patients treated with any benzodiazepine at least for 4 weeks on a stable dose.
* Hamilton Anxiety Rating Scale score major or equal to 20 and a score major or equal to 2 on items 1 and 2 of the same scale at both screening and baseline.
* Clinical Global Impression-Severity major or equal to 4 at both screening and baseline.

Exclusion Criteria:

* Unable to give informed consent.
* Currently participating in another clinical research.
* Any other psychiatric disorder not included in the Anxiety Disorders section of the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-V). Secondary diagnosis of other anxiety disorders are allowed provided the diagnosis is not more prominent than generalized anxiety disorder symptoms.
* Suicide risk as assessed by the researcher at screening or baseline.
* History of substance abuse in the previous six months before the screening visit.
* Suffering a medically relevant or instable disease.
* If woman, being pregnant at screening visit.
* If woman, being breastfeeding.
* A score major or equal to 20 on the Montgomery-Asberg Depression Rating Scale at screening or baseline.
* As judged by a researcher, the patient might not adhere to the intervention or complete follow-up.
* History of use of a banned drug in the past two weeks prior the baseline visit; three weeks in the case of monoamine oxidase inhibitors; one week in the case of fluvoxamine or a tricyclic antidepressant; two weeks for any antipsychotic and; six weeks por long-acting injectable antipsychotics.
* History of use of L-glutamine the most part of the days of the previous month before the baseline visit.
* History of psychotherapy treatment in the past month before the baseline visit.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2019-01-18 (Actual); Primary Completion 2020-05-12 (Actual); Study Completion 2020-05-12 (Actual)

PRIMARY OUTCOMES:
Response on Clinical Global Impression-Improvement | Change from baseline to week 8
  Score of 1 or 2

SECONDARY OUTCOMES:
Response on Hamilton Anxiety Rating Scale | Change from baseline to week 8
  Reduction of baseline score major or equal to 50 %
Reduction of Hamilton Anxiety Rating Scale score | Change from baseline to week 8
  Difference between baseline and final score

CONTACTS AND LOCATIONS:
Overall Officials: José A Ontiveros Sánchez De la Barquera, MD, PhD, Study Chair — Hospital Universitario Dr. Jose E. Gonzalez; Luis A Centeno Gándara, MD, Principal Investigator — Hospital Universitario Dr. Jose E. Gonzalez
Locations (1):
- Hospital Universitario Dr. Jose E. Gonzalez, Monterrey, Nuevo León, Mexico